CLINICAL TRIAL: NCT05546671
Title: Usefulness of Hand Grip Strength as a Predictor of Prolonged Hospital Stay in Elderly Patients Undergoing Cardiac Surgery
Brief Title: Impact of Hand Grip Strength on Length of Hospital Stay After Cardiac Surgery Among Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Kartal Kosuyolu High Speciality Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Can Topcu, Cardiovascular Surgery Specialist, Kartal Kosuyolu High Speciality Training and Research Hospital
Other Study IDs: 2022/13/621
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Strong grippers
  Interventions: Diagnostic Test: Hand grip strength measurement
- Weak grippers
  Interventions: Diagnostic Test: Hand grip strength measurement

INTERVENTIONS:
Diagnostic Test: Hand grip strength measurement — Preoperative hand grip strength will be measured in kilograms using a digital hand dynamometer (Baseline Smedley Digital Hand Dynamometer, Model 12-0286, Baseline Evaluation Instruments, China). Participants will be instructed to grip the hand dynamometer for 5 seconds with their dominant hand 3 times. They will be allowed to rest for 20 second between each grip. The highest measurement of 3 attempts will be recorded. Participants will be categorized as "strong grippers" or "weak grippers" according to Fried criteria as previously defined by Linda P. Fried and colleagues. A weak grip will be defined as follows:
  For men:
  BMI ≤24: hand grip strength ≤29 kg; BMI =24.1 to 28: hand grip strength ≤30 kg; BMI >28: hand grip strength ≤32 kg
  For women:
  BMI ≤23: hand grip strength ≤17 kg; BMI =23.1 to 26: hand grip strength ≤17.3 kg; BMI =26.1 to 29: hand grip strength ≤18 kg; BMI >29: hand grip strength ≤21 kg

SUMMARY:
Hand grip strength has been shown to be a predictor of adverse cardiovascular outcomes in the elderly population. This study aims to investigate whether measurement of hand grip strength could be used as a predictor of prolonged hospital stay after cardiac surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Undergoing isolated coronary artery bypass grafting or isolated valve surgery or combined coronary and valve procedures
* Being oriented and cooperative enough to understand and comply with the instruction of gripping the hand dynamometer

Exclusion Criteria:

* Age <70 years
* Emergent status
* Hemodynamic instability
* Inability to cooperate due to neurocognitive disorder
* Loss of upper extremity motor function of any degree (such as due to previous stroke)
* History of upper extremity amputation of any level

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Study population will be comprised of all consecutive patients ≥70 years of age undergoing elective coronary artery bypass and/or valve surgery at the Department of Cardiovascular Surgery at Kosuyolu Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Prolonged hospital stay | 14 days
  Prolonged hospital stay is defined as postoperative hospital stay for ≥14 days.

SECONDARY OUTCOMES:
Prolonged intensive care unit stay | 48 hours
  Prolonged intensive care unit stay is defined as postoperative intensive care unit stay for >48 hours. This includes sum of all time spent in intensive care unit including unplanned returns.
Prolonged mechanical ventilation | 12 hours
  Prolonged mechanical ventilation is defined as mechanical ventilation of >12 hours. This includes re-intubations and non-invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosuyolu High Specialization Education and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Perry IS, Pinto LC, da Silva TK, Vieira SRR, Souza GC. Handgrip Strength in Preoperative Elective Cardiac Surgery Patients and Association With Body Composition and Surgical Risk. Nutr Clin Pract. 2019 Oct;34(5):760-766. doi: 10.1002/ncp.10267. Epub 2019 Mar 13. PMID 30864228
- [Background] Fu L, Zhang Y, Shao B, Liu X, Yuan B, Wang Z, Chen T, Liu Z, Liu X, Guo Q. Perioperative poor grip strength recovery is associated with 30-day complication rate after cardiac surgery discharge in middle-aged and older adults - a prospective observational study. BMC Cardiovasc Disord. 2019 Nov 27;19(1):266. doi: 10.1186/s12872-019-1241-x. PMID 31775633
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156